CLINICAL TRIAL: NCT04322149
Title: A Phase 2a Open-Label, Multi-Center Study to Evaluate the Safety and Tolerability of Multiple Doses of AT-1501 in Adults With ALS
Brief Title: Multiple Doses of AT-1501-A201 in Adults With ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anelixis Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Organization: Eledon Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-1501-A201
Record Dates: First submitted 2020-03-20; First posted 2020-03-26 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's Disease; motor neuron disease; motor neuron degeneration; AT-1501; humanized blocking antibody to CD40LG; CD40L inhibitor; monoclonal antibody
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AT-1501 (Experimental): 4 sequential dose cohorts
  Interventions: Drug: AT-1501

INTERVENTIONS:
Drug: AT-1501 — AT-1501 monoclonal antibody targeting CD40L given as an IV infusion

SUMMARY:
This is a Phase 2a, multi-center, open label, multiple dose study of AT-1501, a humanized monoclonal antibody antagonist to CD40 ligand (CD40L). Approximately 54 adults with Amyotrophic Lateral Sclerosis (ALS) will be enrolled into the study in the United States and Canada at approximately 13 ALS treatment sites.

Participants will be enrolled into one of four ascending doses.

DETAILED DESCRIPTION:
This is a Phase 2a, multi-center, open label, multiple dose study of AT-1501, a humanized monoclonal antibody antagonist to CD40L. Approximately 54 adults with ALS will be enrolled into the study in the United States and Canada at approximately 13 ALS treatment sites.

Four ascending doses of AT-1501 will be administered as an IV infusion to sequentially enrolling cohorts. Each participant will receive 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.

The study is estimated to take 19 weeks for participants.

ELIGIBILITY:
Inclusion Criteria:

1. ALS diagnosed as possible, laboratory supported probable, probable, or definite as defined by revised El Escorial criteria
2. ALS Functional Rating Scale - Revised (ALSFRS-R) Aggregate score of 37 or greater
3. No more than 24 months from diagnosis

Exclusion Criteria:

1. Any other central or peripheral nervous system disease that may interfere with the evaluation of ALS or its progression
2. Presence of a tracheostomy, or use of permanent assistive ventilation (ventilatory support for 23 hours per day or more)
3. History of malignancy within the previous 5 years, except for localized non-melanoma skin cancers
4. Abnormal function of the immune system resulting from:

   * Clinical conditions affecting the immune system (e.g. HIV infection, agammaglobulinemia),
   * Systemic administration of corticosteroids (PO/IV/IM) at a dose equivalent to 20 mg/day of prednisone for more than 14 consecutive days within 90 days prior to screening,
   * Administration of anti-neoplastic and/or immunomodulating agents (e.g. Tumor necrosis factor alpha (TNF α) antagonists or anti-B cell antibodies) or radiotherapy within 1 year prior to screening.
5. Recipient of Stem Cell or Gene Therapy
6. Positive test for Hepatitis B surface antigen, Hepatitis C antibody, or HIV.
7. History of deep venous thrombosis or pulmonary embolism
8. History of active substance abuse within the past 2 years
9. History of stroke, poorly controlled or significant cardiovascular disease, diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Bornstein, MD, Study Chair — Eledon Pharmaceuticals
Locations (13):
- United States (12):
  - Barrows Neurological Institute, Phoenix, Arizona
  - University of California Irvine, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Augusta University, Augusta, Georgia
  - University of Indiana, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hospital for Special Surgery (HSS), New York, New York
  - Providence Brain & Spine Institute, Portland, Oregon
  - Texas Neurology, P.A., Dallas, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
- Montreal Neurological Institute and Hospital, Montreal, Canada

REFERENCES:
- [Derived] Perrin S, Ladha S, Maragakis N, Rivner MH, Katz J, Genge A, Olney N, Lange D, Heitzman D, Bodkin C, Jawdat O, Goyal NA, Bornstein JD, Mak C, Appel SH, Paganoni S. Safety and tolerability of tegoprubart in patients with amyotrophic lateral sclerosis: A Phase 2A clinical trial. PLoS Med. 2024 Oct 31;21(10):e1004469. doi: 10.1371/journal.pmed.1004469. eCollection 2024 Oct. PMID 39480764

RESULTS

PARTICIPANT FLOW:
Groups:
- AT-1501 1.0 mg/kg: This group received a 1.0 mg/kg dose administered as an 1-hour IV infusion. Each participant received 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.
- AT-1501 2.0 mg/kg: This group received a 2.0 mg/kg dose administered as an 1-hour IV infusion. Each participant received 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.
- AT-1501 4.0 mg/kg: This group received a 4.0 mg/kg dose administered as an 1-hour IV infusion. Each participant received 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.
- AT-1501 8.0 mg/kg: This group received a 8.0 mg/kg dose administered as an 1-hour IV infusion. Each participant received 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.
Period: Overall Study
Arm/Group | AT-1501 1.0 mg/kg | AT-1501 2.0 mg/kg | AT-1501 4.0 mg/kg | AT-1501 8.0 mg/kg
Started | 9 | 9 | 18 | 18
Completed | 8 | 7 | 18 | 16
Not Completed | 1 | 2 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Undergoing cancer treatment & was unable to return to site to complete EOS visit within window | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AT-1501 1.0 mg/kg | AT-1501 2.0 mg/kg | AT-1501 4.0 mg/kg | AT-1501 8.0 mg/kg | Total
Number analyzed (Participants) | 9 | 9 | 18 | 18 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 15 | 11 | 39
  >=65 years | 2 | 3 | 3 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (6.5) | 59 (14.76) | 56.4 (8.53) | 60.3 (11.11) | 59 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 6 | 8 | 19
  Male | 6 | 7 | 12 | 10 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 9 | 9 | 18 | 15 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 9 | 8 | 17 | 18 | 52
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
ALSFRS-R Total Score at Screening [Mean (Standard Deviation); unit: units on a scale] — The ALS Functional Rating Scale - Revised (ALSFRS-R) measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. Each function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Function scores are summed to compute the total score.
  units on a scale | 41.1 (3.02) | 40.2 (1.92) | 39.7 (3.69) | 39.2 (2.65) | 39.9 (3.0)
ALSFRS-R Subdomain at Screening [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The ALS Functional Rating Scale - Revised (ALSFRS-R) measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. The functions reported individually for this study are dyspnea, orthopnea, and respiratory insufficiency. The functions are scored from 4 (normal) to 0 (no ability).
  units on a scale
    Dyspnea | 4 (0) | 3.8 (0.44) | 3.7 (0.59) | 3.8 (0.43) | 3.8 (0.46)
    Orthopnea | 4.0 (0) | 3.8 (0.67) | 3.9 (0.32) | 3.9 (0.24) | 3.9 (0.35)
    Respiratory Insufficiency | 4.0 (0) | 4.0 (0) | 3.9 (0.47) | 3.7 (0.57) | 3.9 (0.44)
ALSFRS-R Total Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The ALS Functional Rating Scale - Revised (ALSFRS-R) measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. Each function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Function scores are summed to compute the total score.
  units on a scale | 40.4 (3.17) | 40.0 (2.0) | 39.6 (3.99) | 38.6 (3.96) | 39.5 (3.56)
ALSFRS-R Subdomain at Baseline [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The ALS Functional Rating Scale - Revised (ALSFRS-R) measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. The functions reported individually for this study are dyspnea, orthopnea, and respiratory insufficiency. The functions are scored from 4 (normal) to 0 (no ability).
  units on a scale
    Dyspnea | 4.0 (0) | 3.7 (0.50) | 3.6 (0.85) | 3.8 (0.55) | 3.7 (0.62)
    Orthopnea | 4.0 (0) | 3.8 (0.67) | 3.8 (0.38) | 3.9 (0.24) | 3.9 (0.37)
    Respiratory Insufficiency | 4.0 (0) | 4.0 (0) | 3.9 (0.47) | 3.7 (0.59) | 3.9 (0.45)
Time Since ALS Symptom Onset [Mean (Standard Deviation); unit: days] | 610.2 (340.20) | 647.2 (388.67) | 705.0 (580.30) | 631.4 (431.02) | 655.1 (457.45)
Time Since ALS Diagnosis [Mean (Standard Deviation); unit: days] | 251.9 (241.52) | 101.6 (75.32) | 244.8 (204.40) | 219.1 (174.57) | 231.5 (188.57)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Incidence of adverse events (AEs) reported as number of participants with at least one TEAE (Treatment Emergent Adverse Event) and at least one SAE (Serious Adverse Event).
Time Frame: Up to 18 Weeks
Population: Full analysis set. All enrolled patients.
Measure: Number; unit: participants
Groups:
- AT-1501 2.0 mg/kg: administered as an 1-hour IV infusion. Each participant received 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.
  This group received a 2.0 mg/kg dose administered as an 1-hour IV infusion. Each participant received 6 bi-weekly (every other week) infusions of AT-1501 over an 11-week period.
Arm/Group | AT-1501 1.0 mg/kg | AT-1501 2.0 mg/kg | AT-1501 4.0 mg/kg | AT-1501 8.0 mg/kg
Number analyzed (Participants) | 9 | 9 | 18 | 18
participants
  Number of Subjects with at Least One TEAE | 8 | 8 | 10 | 16
  Number of Subjects with at Least One SAE | 0 | 1 | 0 | 0

2. Primary Outcome: Safety and Tolerability
Description: Incidence of adverse events (AEs) reported as number of TEAEs (Treatment Emergent Adverse Events) having occurred.
Time Frame: Up to 18 Weeks
Population: Full analysis set. All enrolled patients.
Measure: Number; unit: TEAEs
Arm/Group | AT-1501 1.0 mg/kg | AT-1501 2.0 mg/kg | AT-1501 4.0 mg/kg | AT-1501 8.0 mg/kg
Number analyzed (Participants) | 9 | 9 | 18 | 18
TEAEs | 30 | 66 | 54 | 67

ADVERSE EVENTS:
Time Frame: All serious adverse events were collected from the time of informed consent to 4 weeks after a patient's last dose of investigational product. All adverse events were collected from the first administration of investigational product until completion of the final visit, up to 15 weeks.
Arm/Group | AT-1501 1.0 mg/kg | AT-1501 2.0 mg/kg | AT-1501 4.0 mg/kg | AT-1501 8.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/9 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 8/9 | 8/9 | 10/18 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AT-1501 1.0 mg/kg (N=9) | AT-1501 2.0 mg/kg (N=9) | AT-1501 4.0 mg/kg (N=18) | AT-1501 8.0 mg/kg (N=18)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AT-1501 1.0 mg/kg (N=9) | AT-1501 2.0 mg/kg (N=9) | AT-1501 4.0 mg/kg (N=18) | AT-1501 8.0 mg/kg (N=18)
Headache (Nervous system disorders) | 3 | 2 | 3 | 3
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 4 | 3 | 0 | 7
Asthenia (General disorders) | 0 | 1 | 0 | 1
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0
Feeling jittery (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 5 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Extra-axial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0 | 1
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 3
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI will not submit any results of the Study until after the first to occur: publication of the trial results, notification by Sponsor the trial submission is no longer planned, or the 18 month anniversary of the completion or early termination of the trial. A copy of any proposed publication or disclosure of the results of the Study will be given to Sponsor for review at least 30 days prior to the date of submission for publication (including abstracts) or of public disclosure

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT04322149/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04322149/SAP_001.pdf